CLINICAL TRIAL: NCT03067259
Title: Impact of Anesthesia Surgical Procedure on the Development of Long-term Cognitive Dysfunction
Brief Title: Post Operative Cognitive Dysfunction
Acronym: POCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, FRANCISCO CARLOS BONOFIGLIO, Anesthesiology Doctor, Hospital Italiano de Buenos Aires
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2813
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Complications
Keywords: eldery patients; cognitive impairment
MeSH Terms: conditions — Postoperative Complications; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): It comprises patients who will not undergo any surgical / anesthetic act
- Exposure Group (Other): It comprises those patients that will undergo sedation for diagnostic procedure or some surgical / anesthetic process
  Interventions: Other: Exposure Group

INTERVENTIONS:
Other: Exposure Group — Surgeries of high or low impact. They could be local , regional o general anesthesia; sedation or a combination of both.
  Arms: Exposure Group

SUMMARY:
The objective of this study will be to estimate the incidence of postoperative cognitive dysfunction (DCPO) in patients over 65 years of age, undergoing surgical / anesthetic procedures and in patients who will not undergo surgical / anesthetic. The patients will be taken from the Hospital Italiano de Buenos Aires.

DETAILED DESCRIPTION:
Prospective Study The objective of this study will be to estimate the incidence of Post Operative Cognitive Dysfunction (POCD) in patients over 65 years of age, undergoing surgical / anesthetic procedures and in patients who will not undergo surgical / anesthetic. The patients will be taken from the Hospital Italiano de Buenos Aires.

The population of the present study will be constituted by patients belonging to the HIBA Health Plan. It comprises patients who will not undergo any surgical / anesthetic act (Control Group) and those who will undergo sedation for diagnostic procedure or some surgical / anesthetic process (Exposure Group).

All patients will be tested, the day of signing the Informed Consent (IC), which will serve as an exclusion criterion.

Patients in the Exposure Group who signed the consent will be evaluated on five occasions: up to the day before the surgical / anesthetic act, on the day of the surgical / anesthetic event, 7 days (CAM - If the patient is hospitalized this test will do the test personally if the patient is discharged, the test will be done by telephone), 3 months later and a year after the procedure (for the latter two patients will be asked to attend the Hospital in time). Trained and trained personnel will be in charge of taking the test (which last approximately 1 hour). The battery of tests (detailed below) aims to determine if there is a cognitive decline, to estimate and compare it among the participants of this study.

Patients in the control group will be evaluated on 2 occasions only, a first evaluation on the day the patient and the researchers arrange and then, 12 months from that date.

ELIGIBILITY:
Inclusion Criteria:

or surgical / anesthetic and sedation.

* Patients who have not been exposed in the last 12 months to any of the cases mentioned above.
* Patients with scheduled surgeries will be included, both in the outpatient clinic and with requirements for hospitalization in the floor or in closed units (ICU, UC, etc.), and patients with diagnostic studies or therapeutic procedures requiring anesthesia for their performance by the other.
* Patients will be included with absence of anesthetic or surgical / anesthetic act and sedation in the last 12 months.
* Patients with complete primary schooling (6 years) will be included.

Exclusion Criteria:

* Negative to participate or manage Informed Consent
* MoCa (≤ 26)
* Previous diagnosis of dementia
* Psychosis
* Depression. (GDS Yesavage> 5)
* Toxic Substance abuse of Alcohol according to DSM4 Psychoactive Substances.

  • Use of Illicit drug
* The presence of any congenital or acquired disease or injury that could generate cognitive deficit. (Whether psychiatric, neurological, or metabolic)
* Previous neurosurgery.
* Language barriers.
* Decreased marked visual or auditory acuity that enable from performing the study tests.
* Patients receiving antipsychotics, opioids, anticholinergics or patients who may have varied the benzodiazepines doze or other psychoactive drugs in the last 30 days.
* Patient with cancer disease and life expectancy less than 1 year ( patients will be evaluated from the medical point of view from the records of clinical history according to tumor type, extent,etc.)
* Patients undergoing emergency surgery.
* Patients who have received anesthesia in the past 12 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Estimate the incidence of Post Operative Cognitive Dysfunction (POCD) | 1 year
  We will measure the cognitive impairment using a battery of cognitive tests .
Estimate the incidence of Post Operative Cognitive Dysfunction (POCD) | 1 year
  Check the differences at 12 months after starting the study.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco FB Bonofiglio, PHD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BEDFORD PD. Adverse cerebral effects of anaesthesia on old people. Lancet. 1955 Aug 6;269(6884):259-63. doi: 10.1016/s0140-6736(55)92689-1. No abstract available. PMID 13243706
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] Hudetz JA, Iqbal Z, Gandhi SD, Patterson KM, Hyde TF, Reddy DM, Hudetz AG, Warltier DC. Postoperative cognitive dysfunction in older patients with a history of alcohol abuse. Anesthesiology. 2007 Mar;106(3):423-30. doi: 10.1097/00000542-200703000-00005. PMID 17325499
- [Background] Price CC, Garvan CW, Monk TG. Type and severity of cognitive decline in older adults after noncardiac surgery. Anesthesiology. 2008 Jan;108(1):8-17. doi: 10.1097/01.anes.0000296072.02527.18. PMID 18156877
- [Background] Rasmussen LS. Postoperative cognitive dysfunction: incidence and prevention. Best Pract Res Clin Anaesthesiol. 2006 Jun;20(2):315-30. doi: 10.1016/j.bpa.2005.10.011. PMID 16850780
- [Background] Spiegel DR, Chen V. A case of postoperative cognitive decline, with a highly elevated C- reactive protein, status post left ventricular assist device insertion: a review of the neuroinflammatory hypothesis of delirium. Innov Clin Neurosci. 2012 Jan;9(1):35-41. PMID 22347689
- [Background] Krenk L, Rasmussen LS. Postoperative delirium and postoperative cognitive dysfunction in the elderly - what are the differences? Minerva Anestesiol. 2011 Jul;77(7):742-9. PMID 21709661